CLINICAL TRIAL: NCT01324713
Title: Does Gender Play a Role in Bone-mineral Density Measurement Precision?
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2010-1075
Record Dates: First submitted 2010-09-30; First posted 2011-03-29 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Males
- Females

SUMMARY:
Bone mineral density (BMD) measurement using dual-energy x-ray absorptiometry (DXA) is the current gold standard for osteoporosis diagnosis and therapy monitoring. Like all quantitative tests, there is some variability in BMD results obtained when scanning a person more than once. As such, it is current clinical practice, based on the recommendation of the International Society for Clinical Densitometry, that each technologist perform a precision assessment. This approach consists of scanning 30 people twice; the data from which allow determination of what constitutes a real difference in BMD with 95% confidence. A precision assessment typically evaluates a specific clinic's population, using the age range and genders seen at that clinic. However men generally have larger, but often more arthritic, bones than women which may impact the precision results. Therefore, it is possible that gender-specific precision values should be used in clinical practice, however this issue has never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Able and willing to sign informed consent

Exclusion Criteria:

* Inability to have DXA scans performed due to weight ≥ 450 pounds (exceeds densitometer table limit)
* Metallic hardware in, or overlaying, any of the measured skeletal sites

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population will consist of 90 men and 90 women volunteers who are aged 65 years and older, able and willing to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
DXA Bone Mineral Density precision | 1 day
  The primary analysis will compare DXA BMD precision (mean square error/variance) in males and females, pooled across technicians, using the two-sample F-test for equality of variances. Separate analyses will also be performed for each technician. In addition, due to the sensitivity of the F-test to the normality assumption, a secondary analysis will perform the same comparisons using Levene's test. A nominal two-sided p-value of 0.05 will be regarded as statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Osteoporosis Clinical Center and Research Program, Madison, Wisconsin, United States